CLINICAL TRIAL: NCT06837844
Title: Combined Intrathecal Dexmedetomidine and Adductor Canal Block for Analgesia After Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Combined Intrathecal Dexmedetomidine and Adductor Canal Block for Analgesia After Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Sherif Kamal Arafa, Assistant Professor of Anesthesiology, Surgical Intensive Care and Pain Management Department, Faculty of Medicine, KafrElsheikh University, KafrElsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 50-1-7
Record Dates: First submitted 2025-02-13; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Intrathecal Dexmedetomidine; Adductor Canal Block; Analgesia; Total Knee Arthroplasty
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group ITD (Experimental): Patients will receive 15mg in 3ml hyperbaric bupivacaine intrathecally with 5 μg in 0.5ml dexmedetomidine + adductor canal block using 20 ml saline 0.9% at the end of surgery
  Interventions: Drug: Intrathecal Dexmedetomidine
- Group ACB (Active Comparator): Patients will receive 15mg in 3ml hyperbaric bupivacaine intrathecally with 0.5ml saline 0.9% + adductor canal block using 20 ml bupivacaine 0.25% at the end of surgery.
  Interventions: Drug: Adductor Canal Block
- Group ITD+ACB (Experimental): Patients will receive 15mg in 3ml hyperbaric bupivacaine intrathecally with 5 μg in 0.5ml dexmedetomidine + adductor canal block using 20 ml bupivacaine 0.25% at the end of surgery.
  Interventions: Drug: Intrathecal Dexmedetomidine + Adductor Canal Block

INTERVENTIONS:
Drug: Intrathecal Dexmedetomidine — Patients will receive 15mg in 3ml hyperbaric bupivacaine intrathecally with 5 μg in 0.5ml dexmedetomidine + adductor canal block using 20 ml saline 0.9% at the end of surgery
  Arms: Group ITD
Drug: Adductor Canal Block — Patients will receive 15mg in 3ml hyperbaric bupivacaine intrathecally with 0.5ml saline 0.9% + adductor canal block using 20 ml bupivacaine 0.25% at the end of surgery.
  Arms: Group ACB
Drug: Intrathecal Dexmedetomidine + Adductor Canal Block — Patients will receive 15mg in 3ml hyperbaric bupivacaine intrathecally with 5 μg in 0.5ml dexmedetomidine + adductor canal block using 20 ml bupivacaine 0.25% at the end of surgery.
  Arms: Group ITD+ACB

SUMMARY:
The aim of this work is to evaluate the effect of combined intrathecal dexmedetomidine and adductor canal block for analgesia after total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Effective postoperative pain management is essential for improving patient outcomes following knee surgery, facilitating early mobilization, and reducing the risk of complications.

The adductor canal block (ACB) is a nerve block of Hunters canal, which includes the saphenous and vastus medialis nerves. Additionally, other sensory nerves, such as the femoral nerve, medial cutaneous nerve, and both the anterior branch and terminal end of the posterior branch of the obturator nerve to some extent as it enters the distal part of the canal are blocked by the ACB.

Dexmedetomidine (DXM) a highly selective α2 adrenergic agonist with sedative, anxiolytic, analgesic, sympatholytic and antihypertensive effects.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for total knee arthroplasty under spinal anesthesia.

Exclusion Criteria:

* Patients with neurological or intellectual disability.
* History of allergy to local anesthetics or dexmedetomidine .
* Infection at the injection site.
* Prolonged use of analgesic or sedative medications.
* Coagulation abnormalities.
* Pregnancy.
* Obesity [body mass index (BMI) > 30 kg/m2].

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 48 hours postoperatively
  The patient will receive a 3mg bolus of morphine as a rescue analgesic if the visual analog scale (VAS) was greater than 3, and if the pain persisted for more than 30 mins, the injection was repeated until the VAS became below 4

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperatively
  Time to the 1st rescue analgesia will be recorded from the end of surgery till the first dose of morphine administered.
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analog scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively
Heart rate | In post-anesthesia care unit (PACU) (Up to 1 hour)
  Heart rate will be recorded every 5 minutes till the end of surgery and in post-anesthesia care unit (PACU).
Mean arterial pressure | In post-anesthesia care unit (PACU) (Up to 1 hour)
  Mean arterial pressure will be recorded every 5 minutes till the end of surgery and in post-anesthesia care unit (PACU).
Degree of patient satisfaction | 48 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of adverse events | 48 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.